CLINICAL TRIAL: NCT01602042
Title: Phase II Study: Adaptive Portable Essential Tremor Monitor
Brief Title: Adaptive Portable Essential Tremor Monitor
Status: Completed | Type: Observational
Sponsor: Great Lakes NeuroTechnologies Inc. (Industry)
Collaborators: Rush University Medical Center (Other); Baylor College of Medicine (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2R44AG034708-02A1 (NIH)
Record Dates: First submitted 2012-05-16; First posted 2012-05-18 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-12

CONDITIONS: Essential Tremor
Keywords: essential tremor; motion sensors; tremor
MeSH Terms: conditions — Essential Tremor; Tremor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to evaluate the utility of a portable motion sensor-based system designed to monitor essential tremor (ET) to better prescribe therapy to minimize symptoms and expand care for ET patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Clinical diagnosis of essential tremor
* Able to provide informed consent

Exclusion Criteria:

* Significant medical or psychiatric illness
* Not capable of following the required clinical instructions
* Serious medical conditions that compromise safety

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Essential tremor
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2012-05; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Tremor ratings during activities of daily living versus standardized tasks. | 10 hours each day the sensor is worn.

CONTACTS AND LOCATIONS:
Overall Officials: Dustin A Heldman, PhD, Principal Investigator — CleveMed Inc. also dba Great Lakes NeuroTechnologies
Locations (2):
- United States (2):
  - Rush University Medical Center, Chicago, Illinois
  - Baylor College of Medicine, Houston, Texas